CLINICAL TRIAL: NCT01863108
Title: Dose-escalation Study to Assess the Safety and Tolerability of Sub-cutaneous Injections of a Peptide-loaded Plasmacytoid Dendritic Cell Line (GeniusVac-Mel4) in Patients With Melanoma
Brief Title: Safety Study of a Dendritic Cell-based Cancer Vaccine in Melanoma
Acronym: GeniusVac-Mel4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Etablissement Français du Sang (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Joseph Fourier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 11 19; 2012-003124-20 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Tumor Vaccines; Effects of Immunotherapy
Keywords: Melanoma; Immunotherapy; Dermatology; cancer vaccine; Plasmacytoid dendritic cell line; Advanced Medicinal Therapy Product; allogeneic
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GeniusVac-Mel4 (Experimental): Sub-cutaneous injections of GeniusVac-Mel4 in patients with melanoma.
  Interventions: Biological: GeniusVac-Mel4

INTERVENTIONS:
Biological: GeniusVac-Mel4 — Multiple sub-cutaneous injections (1 injection weekly during 3 weeks) of GeniusVac-Mel4 (3 increasing dose groups) in patients with melanoma

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple sub-cutaneous injections of GeniusVac-Mel4, a dendritic cell-based cancer vaccine, in patients with melanoma. The secondary objectives are to determine immune response and clinical efficacy of such injections in patients with melanoma.

DETAILED DESCRIPTION:
GeniusVac-Mel4 is a drug product composed of an irradiated allogeneic plasmacytoid dendritic cell (PDC) line loaded with 4 melanoma peptides derived from Melan-A, gp100, Tyrosinase or Mage-A3. This cell line is HLA-A*02:01, a phenotype found in 40% of the European population. This approach exploits the PDC line high capacity of boosting anti-tumor cytotoxic response against melanoma antigens in HLA-A*02:01 melanoma patients. In the preclinical studies, a strong proof of concept was brought. Indeed, the GeniusVac-Mel4 capacity to induce high number of cytotoxic antitumor T-cells was shown in melanoma model, both in vivo in humanized mice and ex vivo with patients' PBMC (peripheral blood mononuclear cells) (Aspord et al 2010 and 2012).

It is planned to include patients in three dose-escalating groups (4, 20, 60 millions of GeniusVac-Mel4 cells). At least, 3 patients will be recruited in each dose group of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic melanoma (at stage IIIC or stage IV under the AJCC 2009 classification not surgically resectable.
* Patients who do not respond to at least one line of systemic treatment
* Male and female (with β-HCG negative test)
* Patients HLA-A*0201
* Age > 18 years
* Blood parameters (Hemoglobin ≥ 10g/dl, Leucocytes ≥ 4000/μl,Lymphocytes ≥ 1000/μl, Platelets ≥100.000/μl, creatinin ≤ 2.0mg/dl, bilirubin ≤ 2.0mg/dl, ASAT and ALAT ≤ 2.5 fold the upper normal level)
* OMS performance score < 3
* Informed written consent.

Exclusion Criteria:

* Positive serology for HCV, HTLV, HIV, active hepatitis
* Protected persons according to French regulations articles L1121-5 to L1121-8 (Public Health Code)
* Non-pregnant women without effective contraception
* Any serious acute or chronic illness, for example: active infection, coagulation disorder.
* Presence of a second cancer in the 5 years preceding inclusion into the study with the exception of in situ cervical carcinoma or a cutaneous carcinoma or other melanoma.
* Intercurrent disease requiring corticosteroids.
* Any active autoimmune disease including insulin dependent diabetes mellitus. Vitiligo or autoimmune thyroid disease are not criteria for exclusion.
* Autoimmune eye disease.
* Evidence of immunosuppression for any reason
* Primary ocular melanoma
* Chemotherapy, immunotherapy or radiotherapy in the 4 weeks preceding inclusion (6 weeks in the case of nitroso-urea and mitomycin C).
* Treatment with drugs under development within 4 weeks.
* Cerebral metastases metastasis with the exception of: known metastasis previously treated by surgery or stereotactic radio-surgery, AND Cerebral metastasis, if still present, must be stable for at least 90 days before inclusion and documented with two consecutive MRI or scanner with contrast media, AND, asymptomatic
* Existence of any surgical or medical condition which, in the judgment of the Investigator, might interfere with this study.
* Patients who are not willing to comply with the provisions of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06; Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of a multiple sub-cutaneous injections of GeniusVac-Mel4. | 1 year
  Safety and tolerance is monitored by performing clinical laboratory tests, assessments of vital signs, full clinical examination, occurrence of adverse events.

SECONDARY OUTCOMES:
Evaluation of the immune response | 1 year
  The induction of an immune response is evaluated at several time points by measuring :
  * The frequency of the T lymphocytes specific for each peptide used in the protocol.
  * The functionality of these T-cells (cytotoxicity and IFN-g secretion)
Evaluation of the clinical response | 1 year
  The evolution of the disease will be determined with a clinical examination and scanner exams. The overall tumor response will be evaluated in accordance RECIST 1.1 and immune-related response criteria (irRC).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Plumas, PhD, Study Director — Etablissement Français du Sang/Grenoble University/ INSERM U823; Julie Charles, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Aspord C, Leccia MT, Salameire D, Laurin D, Chaperot L, Charles J, Plumas J. HLA-A(*)0201(+) plasmacytoid dendritic cells provide a cell-based immunotherapy for melanoma patients. J Invest Dermatol. 2012 Oct;132(10):2395-2406. doi: 10.1038/jid.2012.152. Epub 2012 Jun 14. PMID 22696054
- [Background] Aspord C, Charles J, Leccia MT, Laurin D, Richard MJ, Chaperot L, Plumas J. A novel cancer vaccine strategy based on HLA-A*0201 matched allogeneic plasmacytoid dendritic cells. PLoS One. 2010 May 4;5(5):e10458. doi: 10.1371/journal.pone.0010458. PMID 20454561
- [Result] Charles J, Chaperot L, Hannani D, Bruder Costa J, Templier I, Trabelsi S, Gil H, Moisan A, Persoons V, Hegelhofer H, Schir E, Quesada JL, Mendoza C, Aspord C, Manches O, Coulie PG, Khammari A, Dreno B, Leccia MT, Plumas J. An innovative plasmacytoid dendritic cell line-based cancer vaccine primes and expands antitumor T-cells in melanoma patients in a first-in-human trial. Oncoimmunology. 2020 Apr 12;9(1):1738812. doi: 10.1080/2162402X.2020.1738812. eCollection 2020. PMID 32313721